CLINICAL TRIAL: NCT00946049
Title: Oral Bacteria on Suture Materials - Clinical Comparison of an Antibacterial-coated and a Non-coated Suture Material (VICRYL PLUS® vs. VICRYL®, Ethicon) in Intraoral Dentoalveolar Surgery
Brief Title: Oral Bacteria on Suture Materials - Clinical Comparison of an Antibacterial-coated and a Non-coated Suture Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Purpose: Treatment
Other Study IDs: 323/05
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Bacterial Colonization
Keywords: Checking clinical antibacterial effect of Vicryl Plus compared to conventional Vicryl in intraoral surgery; Bacteria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vicryl Plus (Experimental)
  Interventions: Device: Vicryl Plus
- Vicryl (Active Comparator)
  Interventions: Device: Vicryl

INTERVENTIONS:
Device: Vicryl Plus
  Arms: Vicryl Plus
Device: Vicryl
  Arms: Vicryl

SUMMARY:
Antibacterial Triclosan-coated suture material (VICRYL PLUS®, Ethicon) and non-coated (VICRYL®) was compared for bacterial colonization after third molar extraction. Sutures were removed postoperatively and adhered bacteria were investigated.

ELIGIBILITY:
Inclusion Criteria:

* planned surgical extraction of 1 to 4 wisdom teeth
* no inflammation and pain within the planned surgical area
* legal age
* clinically healthy patient

Exclusion Criteria:

* allergy to Triclosan or phenols
* gravidity/lactation
* immunosuppression due to drugs or diseases
* severe general diseases
* long-term medication
* intake or use of other antibiotical drugs/devices

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2005-03; Primary Completion 2007-06 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Albert-Ludwigs-University Freiburg, Department for Oral and Maxillofacial Surgery, Freiburg im Breisgau, Germany